CLINICAL TRIAL: NCT03361228
Title: An Open-Label, Multicenter, Nonrandomized, Dose-Escalation, and Tumor-Expansion Phase 1/2 Study to Evaluate the Safety, Tolerability, and Antitumor Activity of INCB001158 Plus Epacadostat (INCB024360), With or Without Pembrolizumab, in Subjects With Advanced Solid Tumors
Brief Title: A Study to Evaluate the Safety, Tolerability, and Antitumor Activity of INCB001158 Plus Epacadostat, With or Without Pembrolizumab, in Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was terminated early based on emerging data with epacadostat and pembrolizumab.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 01158-202
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Results first posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Solid Tumors
Keywords: Non-small cell lung cancer (NSCLC); melanoma; urothelial carcinoma; squamous cell carcinoma of the head and neck (SCCHN); small cell lung cancer (SCLC); colorectal cancer (CRC); arginase 1 inhibitor; indoleamine 2,3-dioxygenase 1 inhibitor; programmed death-1 receptor (PD-1) inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Carcinoma, Transitional Cell; Squamous Cell Carcinoma of Head and Neck; Small Cell Lung Carcinoma; Colorectal Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — epacadostat; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- INCB001158 + Epacadostat + Pembrolizumab (Experimental)
  Interventions: Drug: INCB001158; Drug: Epacadostat; Drug: Pembrolizumab
- INCB001158 + Epacadostat (Experimental)
  Interventions: Drug: INCB001158; Drug: Epacadostat

INTERVENTIONS:
Drug: INCB001158 — Phase 1: INCB001158 administered orally twice daily at the protocol-defined dose. Phase 2: INCB001158 administered orally twice daily at the recommended dose from Phase 1.
Drug: Epacadostat — Epacadostat at the protocol-defined dose administered orally twice daily.
  Other Names: INCB024360
Drug: Pembrolizumab — Pembrolizumab at the protocol-defined dose administered intravenously every 3 weeks.
  Other Names: MK-3475
  Arms: INCB001158 + Epacadostat + Pembrolizumab

SUMMARY:
The purpose of this study is to assess the safety and antitumor activity of INCB001158 plus epacadostat, with or without pembrolizumab, in participants with advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* For Phase 1, subjects with histologically or cytologically confirmed advanced or metastatic solid tumors that have failed prior standard therapy (disease progression; subject intolerance is also allowable).
* For Phase 2, subjects with the following tumor types who meet protocol-defined criteria: advanced or metastatic NSCLC, melanoma, urothelial carcinoma, SCCHN, SCLC, and CRC.
* Presence of at least 1 measurable lesion by computed tomography or magnetic resonance imaging per RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.
* Resolution of all toxicities and any toxic effect(s) of the most recent prior therapy to Grade 1 or less (except alopecia). Subjects with ≤ Grade 2 neuropathy are an exception and may enroll.
* Adequate renal, hepatic, and hematologic functions per protocol-defined laboratory parameters within ≤ 7 days before treatment initiation.

Exclusion Criteria:

* Participation in any other study in which receipt of an investigational study drug or device occurred within 2 weeks or 5 half-lives (whichever is longer) before first dose.
* Has received a prior monoclonal antibody within 4 weeks or 5 half-lives (whichever is shorter) before administration of study drug.
* Prior chemotherapy or targeted small molecule therapy within 2 weeks before administration of study treatment.
* Prior therapy with an IDO1 or arginase 1 inhibitor.
* Active autoimmune disease that has required systemic treatment in past 2 years. Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Receipt of a live vaccine within 30 days before the first dose of study treatment.
* Any history of serotonin syndrome after receiving serotonergic drugs.
* Use of protocol-defined prior/concomitant therapy.
* Known or suspected defect in the function of the urea cycle.
* History of gastrointestinal condition that may affect drug absorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sven Gogov, MD, Study Director — Incyte Corporation
Locations (2):
- United States (2):
  - University of Alabama, Birmingham, Alabama
  - The University of Chicago Medicine, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 3 different sites in US. A total of 10 patients were screened and 5 patients enrolled in study.
Pre-assignment Details: No patients were analyzed due to insufficient numbers and risk of identifying patient by reporting data on 1 person enrolled in cohort 2
Groups:
- INCB001158 50mg BID+ Epacadostat + Pembrolizumab: INCB001158 dosed at 50mg BID in combination with epacadostat (100 mg BID) and pembrolizumab (200 mg Q3W)
- INCB001158 75 mg BID + Epacadostat + Pembrolizumab: INCB001158 dosed at 75mg BID in combination with epacadostat (100 mg BID)and pembrolizumab (200 mg Q3W)
Period: Overall Study
Arm/Group | INCB001158 50mg BID+ Epacadostat + Pembrolizumab | INCB001158 75 mg BID + Epacadostat + Pembrolizumab
Started | 4 | 1
Completed | 0 | 0
Not Completed | 4 | 1
Not completed — Other | 1 | 1
Not completed — Death | 3 | 0

BASELINE CHARACTERISTICS:
Population: No patients were analyzed due to insufficient numbers and risk of identifying patient by reporting data on 1 person enrolled in cohort 2
Groups:
- Total: Total of all reporting groups
Arm/Group | INCB001158 50mg BID+ Epacadostat + Pembrolizumab | INCB001158 75 mg BID + Epacadostat + Pembrolizumab | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous
Sex: Female, Male [unit: participants]
Race/Ethnicity, Customized [unit: participants]
Race/Ethnicity, Customized [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 Only: Safety and Tolerability of INCB001158 in Combination With Epacadostat ± Pembrolizumab as Assessed by Number of Participants With a Treatment-emergent Adverse Event (TEAE)
Description: TEAE defined as any adverse event either reported for the first time or worsening of a pre-existing event after first dose of study treatment.
Time Frame: Up to approximately 12 months per subject
Population: as for baseline characteristics
Arm/Group | INCB001158 50mg BID+ Epacadostat + Pembrolizumab | INCB001158 75 mg BID + Epacadostat + Pembrolizumab
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Phase 2 Only: Objective Response Rate (ORR) of INCB001158 in Combination With Epacadostat ± Pembrolizumab
Description: Defined as percentage of subjects having a complete response (CR) or partial response (PR) based on investigator assessment per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
Time Frame: Up to approximately 12 months per subject
Population: Data was not collected as no participants were enrolled in Phase 2 of the study
Arm/Group | INCB001158 50mg BID+ Epacadostat + Pembrolizumab | INCB001158 75 mg BID + Epacadostat + Pembrolizumab
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Phase 2 Only: Safety and Tolerability of INCB001158 in Combination With Epacadostat ± Pembrolizumab as Assessed by Number of Participants With a TEAE
Description: as for outcome 1
Time Frame: Up to approximately 12 months per subject
Population: Data was not collected as no participants were enrolled in Phase 2 of the study
Arm/Group | INCB001158 50mg BID+ Epacadostat + Pembrolizumab | INCB001158 75 mg BID + Epacadostat + Pembrolizumab
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Phase 1 Only: ORR With INCB001158 in Combination With Epacadostat ± Pembrolizumab
Description: Defined as percentage of subjects having a CR or PR based on investigator assessment per RECIST v1.1.
Time Frame: Up to approximately 12 months per subject
Population: as for baseline characteristics
Arm/Group | INCB001158 50mg BID+ Epacadostat + Pembrolizumab | INCB001158 75 mg BID + Epacadostat + Pembrolizumab
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Disease Control Rate With INCB001158 in Combination With Epacadostat ± Pembrolizumab
Description: Defined as percentage of subjects having CR, PR, or stable disease for at least 56 days based on investigator assessment per RECIST v1.1.
Time Frame: Up to approximately 12 months per subject
Population: as for baseline characteristics
Arm/Group | INCB001158 50mg BID+ Epacadostat + Pembrolizumab | INCB001158 75 mg BID + Epacadostat + Pembrolizumab
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Duration of Response With INCB001158 in Combination With Epacadostat ± Pembrolizumab
Description: Defined as the time from earliest date of disease response until the earliest date of disease progression per RECIST v1.1, or death due to any cause, if occurring sooner than progression.
Time Frame: Up to approximately 12 months per subject
Population: as for baseline characteristics
Arm/Group | INCB001158 50mg BID+ Epacadostat + Pembrolizumab | INCB001158 75 mg BID + Epacadostat + Pembrolizumab
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Progression-free Survival With INCB001158 in Combination With Epacadostat ± Pembrolizumab
Description: Defined as the time from date of first dose of study treatment until the earliest date of disease progression (based on investigator assessment of per RECIST v1.1) or death due to any cause, if occurring sooner than progression.
Time Frame: Up to approximately 12 months per subject
Population: as for baseline characteristics
Arm/Group | INCB001158 50mg BID+ Epacadostat + Pembrolizumab | INCB001158 75 mg BID + Epacadostat + Pembrolizumab
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Plasma Pharmacokinetic Profile of INCB001158 and Epacadostat
Description: Noncompartmental method of analysis will be used to analyze the plasma concentrations of INCB001158 and epacadostat.
Time Frame: Up to approximately 1 month
Population: as for baseline characteristics
Arm/Group | INCB001158 50mg BID+ Epacadostat + Pembrolizumab | INCB001158 75 mg BID + Epacadostat + Pembrolizumab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to approximately 12 months
Description: The safety population included all subjects enrolled in the study who received at least 1 dose of study treatment.
Arm/Group | INCB001158 50mg BID+ Epacadostat + Pembrolizumab | INCB001158 75 mg BID + Epacadostat + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 3/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 3/4 | 1/1
Other Adverse Events (participants affected / at risk) | 4/4 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | INCB001158 50mg BID+ Epacadostat + Pembrolizumab (N=4) | INCB001158 75 mg BID + Epacadostat + Pembrolizumab (N=1)
Myocardial infarction (Cardiac disorders) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | INCB001158 50mg BID+ Epacadostat + Pembrolizumab (N=4) | INCB001158 75 mg BID + Epacadostat + Pembrolizumab (N=1)
Dry eye (Eye disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Oral herpes (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Weight increased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT03361228/Prot_SAP_000.pdf